CLINICAL TRIAL: NCT03202823
Title: Arachidonic Acid Metabolism in Carotid Stenosis Plaque in Diabetic Patients
Acronym: MASCADI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MENEGAUT 2016
Record Dates: First submitted 2017-06-21; First posted 2017-06-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics
  Interventions: Procedure: blood samples; Procedure: recover samples of atheromatous plaque
- Non-diabetics
  Interventions: Procedure: blood samples; Procedure: recover samples of atheromatous plaque

INTERVENTIONS:
Procedure: blood samples — 3 tubes (5 ml volume) collected during surgery
Procedure: recover samples of atheromatous plaque — a carotid sample collected during surgery

SUMMARY:
Diabetes is associated with an increased risk of cardiovascular complications, as a reflection of the chronic inflammatory status. Monocytes-macrophages in diabetic subjects present impaired arachidonic acid metabolism. Moreover, atheromatous plaques in diabetic subjects seem to be significantly enriched in 2-AA-LPC (2-arachidonoyl-lysophosphatidylcholine) and are more inflammatory and more likely to rupture than are plaques in non-diabetic subjects. We therefore hypothesize that this vulnerability of atheromatous plaques in diabetic subjects could be explained by impaired 2-AA-LPC metabolism within the plaque.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided explicit consent
* Patients older than 18 years
* Patients about to undergo surgery for carotid stenosis
* Haemoglobin ≥ 7g/dl at the time the sample is taken
* Respect the maximum volume of blood taken (treatment + research) in 30 days

SPECIFIC TO DIABETICS

- Patients with type 1 or 2 diabetes diagnosed more than 6 months earlier

Exclusion Criteria:

* Patients under guardianship
* Patients without health insurance cover
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and non-diabetic patients with carotid stenosis who undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Change in arachidonic acid metabolism of atheromatous plaques from diabetic versus non-diabetic subjects | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Menegaut L, Laubriet A, Crespy V, Leleu D, Pilot T, Van Dongen K, de Barros JP, Gautier T, Petit JM, Thomas C, Nguyen M, Steinmetz E, Masson D. Inflammation and oxidative stress markers in type 2 diabetes patients with Advanced Carotid atherosclerosis. Cardiovasc Diabetol. 2023 Sep 14;22(1):248. doi: 10.1186/s12933-023-01979-1. PMID 37710315